CLINICAL TRIAL: NCT00585702
Title: Antimanic Drug Use in Pregnancy
Acronym: AMUP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Wisner, Professor of Psychiatry, University of Pittsburgh
Other Study IDs: 1R01MH075921 (NIH); 1R01MH075921 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-03 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Bipolar Disorder; Pregnancy
Keywords: Bipolar Disorder; Pregnancy; Infant Development
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Pregnant women with bipolar disorder
- 2: Pregnant women without bipolar disorder

SUMMARY:
The purpose of this study is to learn about the effects of bipolar disorder or the use of antimanic medications on the mother's health and wellbeing during pregnancy and for the first postpartum year. Infant health and development are also assessed during the first year. Participation in the study includes 7 study visits, three in pregnancy and four postpartum.

ELIGIBILITY:
Inclusion Criteria for Bipolar Subjects:

* Age 18 or older
* Pregnant at 20 weeks or more
* Women must receive OB care
* English-speaking
* DSM-IV diagnosis of BP, any subtype

Inclusion Criteria for non-Bipolar Control Subject:

* Age 18 or older
* Pregnant at 20 weeks or more
* English-speaking
* Women must receive OB care.
* Women may have past or present subclinical Major Depressive Disorder according to the DSM-IV.

Exclusion Criteria for all:

* Women must have no Active Alcohol Abuse or Dependence, Active Abuse or Dependence of Opiates, Inhalants, Amphetamines including Ecstasy or LSD, Active IV Drug Abuse, or Methadone Maintenance.
* Women must not take drugs in the FDA categories D or X.

Additional Exclusion Criteria for Control Subjects:

* Women must have no lifetime history of Bipolar Disorder or antimanic drug use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Age 18 or older Pregnant at 20 weeks or more English-speaking DSM-IV diagnosis of BP, any subtype
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2006-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
SIGH-ADS | 20, 30 36 weeks gestation, 2,12,28,52 weeks postpartum
Mania Rating Scale | 20, 30 36 weeks gestation, 2,12,28,52 weeks postpartum
Bayley Scales of Infant Development | 12, 28, 52 weeks postpartum

SECONDARY OUTCOMES:
Weight gain in pregnancy | 20,30,36 weeks gestation
Structured Clinical Interview for DSM-IV | 20 weeks gestation at enrollment
Nutritional Blood Levels | 20, 30 36 weeks gestation, 2,12,28,52 weeks postpartum
Maternal Functioning and Gratification | 2, 12, 28, 52 weeks postpartum
Infant physical exam | 2,12,28,52 weeks post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Wisner, MD MS, Principal Investigator — Department of Psychiatry, School of Medicine, University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Wisner KL, Sit D, O'Shea K, Bogen DL, Clark CT, Pinheiro E, Yang A, Ciolino JD. Bipolar disorder and psychotropic medication: Impact on pregnancy and neonatal outcomes. J Affect Disord. 2019 Jan 15;243:220-225. doi: 10.1016/j.jad.2018.09.045. Epub 2018 Sep 18. PMID 30248632
- [Derived] Yang A, Ciolino JD, Pinheiro E, Rasmussen-Torvik LJ, Sit DKY, Wisner KL. Neonatal Discontinuation Syndrome in Serotonergic Antidepressant-Exposed Neonates. J Clin Psychiatry. 2017 May;78(5):605-611. doi: 10.4088/JCP.16m11044. PMID 28570796
- [Derived] Santucci AK, Singer LT, Wisniewski SR, Luther JF, Eng HF, Sit DK, Wisner KL. One-Year Developmental Outcomes for Infants of Mothers With Bipolar Disorder. J Clin Psychiatry. 2017 Sep-Oct;78(8):1083-1090. doi: 10.4088/JCP.15m10535. PMID 28068465
- [Derived] Kim DR, Pinheiro E, Luther JF, Eng HF, Dills JL, Wisniewski SR, Wisner KL. Is third trimester serotonin reuptake inhibitor use associated with postpartum hemorrhage? J Psychiatr Res. 2016 Feb;73:79-85. doi: 10.1016/j.jpsychires.2015.11.005. Epub 2015 Nov 19. PMID 26692255